CLINICAL TRIAL: NCT04175639
Title: mHealth Behavioral Cancer Pain Intervention for Medically Undeserved Patients
Brief Title: mHealth Behavioral Cancer Pain Intervention for Medically Underserved Patients
Acronym: ICAN-NC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103527
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: cancer; pain; fatigue; distress; coping; mHealth; symptom management; physical disability
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Pain; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Health Pain Coping Skills Training (mPCST) (Experimental): Mobile Health Pain Coping Skills Training (mPCST) protocol for breast cancer survivors with persistent pain that will produce significant improvements in pain, pain disability, fatigue, physical disability, and adherence to post-treatment lifestyle recommendations that are impacted by pain (i.e., daily activity, self-monitoring of symptoms).
  Interventions: Behavioral: Mobile Health Pain Coping Skills Training (mPCST)
- mHealth-Education (mHealth-Ed) (No Intervention): mHealth-Education (mHealth- Ed): Participating in mHealth will involve four 50-minute individual intervention sessions conducted over the course of 8 weeks with tele-video-conferencing at patient's community-based clinic with a nurse about cancer care.

INTERVENTIONS:
Behavioral: Mobile Health Pain Coping Skills Training (mPCST) — Participating in Mobile Health Pain Coping Skills Training will involve four 50-minute individual intervention sessions conducted over the course of 8 weeks with tele-video-conferencing at patient's community-based clinic. The therapist delivering the intervention will be at Duke University Medical Center, and patients will be at their community clinic.
  Arms: Mobile Health Pain Coping Skills Training (mPCST)

SUMMARY:
The efficacy of a mobile health (mHealth) behavioral cancer pain intervention designed to decrease pain and disability for breast cancer patients in medically underserved areas has not been investigated. The long-term goal of this work is to use mHealth technologies to facilitate wide-spread implementation of an efficacious behavioral cancer pain intervention - a non-pharmacological approach to pain management. The proposed project's objective is to demonstrate the efficacy of an innovative mobile health Pain Coping Skills Training (mPCST-Community) designed to meet the needs of breast cancer patients with pain in medically underserved areas. mPCST-Community addresses intervention barriers for patients in medically underserved areas as it is delivered with video-conferencing in the patients' community based oncology clinic by a remote therapist, is extended to the patients' home environment using simple mHealth technology, and is low-literacy adapted. The central hypothesis is that mPCST-Community will result in decreased pain compared to a mHealth education attention control group (mHealth-Ed). The rationale of this proposal is that if mPCST-Community is shown to be efficacious it will rapidly increase intervention access for individuals who receive their oncology care in medically underserved areas and ultimately reduce pain-related suffering. Guided by strong preliminary data, a randomized controlled trial will be used to pursue three specific aims: 1) Test the extent to which the mPCST-Community intervention reduces pain, fatigue, disability, and distress, 2) Examine self-efficacy and pain catastrophizing as mediators through which the mPCST-Community leads to reductions in pain, fatigue, disability, and distress, and 3) To evaluate the cost-effectiveness of mPCST-Community. For Aim 1, based on the study team's extensive work demonstrating the efficacy of in-person pain coping skills training protocols and pilot work showing promise for mPCST-Community, it is expected that mPCST-Community will lead to decreased pain as well as fatigue, disability, and distress compared to mHealth-Ed. For Aim 2, it is expected that the effects of mPCST-Community will be mediated by increased self-efficacy for pain control and decreased pain catastrophizing. For Aim 3, it is expected that mPCST-Community will demonstrate cost-effectiveness as assessed by all-cause medical resource use, participant and therapist time, and health utilities as well as successful overall accrual, high subject retention, and high intervention adherence.

DETAILED DESCRIPTION:
Guided by extensive prior work, the investigators have designed an innovative mHealth behavioral pain coping skills training (PCST) intervention to reduce pain and disability in cancer patients in medically underserved areas (mPCST-Community). Our prior work has tested PCST protocols through in-person sessions at major medical centers where resources and literacy levels are relatively high. mPCST-Community is different and innovative; it uses mHealth technology (e.g., videoconferencing) to decrease access barriers for patients in medically underserved areas. The protocol is brief (4 sessions) and delivered in the community clinic by a remote well-trained pain therapist. Importantly, this protocol has been carefully adapted for low literacy patients.Beverly Thorn, PhD, a nationally recognized expert in strategies for adapting pain coping interventions to low literacy, medically underserved patients, was instrumental in developing the mPCST-Community protocol. mPCST-Community extends to the patient's daily life through use of a simple mobile application that provides low literacy text/audio protocol summaries, relaxation audio, daily assessment and personalized feedback, and coping messaging.

The investigators propose a randomized controlled trial (RCT) to test the efficacy of the developed mPCST-Community protocol in breast cancer patients with pain receiving cancer care in medically underserved areas (N=180). The investigators have done careful and extensive pilot work to prepare for the proposed trial. Our pilot work (Journal of Psychosocial Oncology) was conducted in breast cancer patients with pain in three medically underserved rural community clinics. First, focus group data (3 groups; n=19) were used to further refine the adapted protocol. Second, the mPCST-Community protocol was evaluated in a single-arm trial with 20 patients. The invesitgators found high feasibility (i.e., recruitment met), low attrition and high adherence (90% completion), and high acceptability. Importantly, impressive and positive pre- to post-intervention changes were found for pain severity (t=-2.52, p=0.01,gav=0.62; 30% change), pain interference (t=-2.62,p=0.01, gav=0.62), and self-efficacy for pain management (t=3.57, p=0.0004, gav=0.98; 30% change).8Study specific aims are:

Aim 1:Test the extent to which mPCST-Community reduces breast cancer patients' pain severity (primary outcome), pain interference, fatigue, physical disability, and psychological distress. Hypothesis:mPCST-Community will lead to decreases in these pain-related outcomes compared to a Health-Ed control condition.

Aim 2:Examine mediators through which mPCST-Community leads to benefits. Hypothesis:The effects of mPCST-Community on pain severity, pain interference, fatigue, physical disability, and psychological distress will be mediated by increased self-efficacy for pain management and decreased pain catastrophizing.

Aim 3:Evaluate the cost and cost-effectiveness of mPCST-Community. Hypothesis: mPCST-Community will be cost-saving or cost effective in terms of its incremental cost per quality-adjusted life-year from a societal perspective, inclusive of healthcare, intervention and patient-time costs. Its sustainability will be further demonstrated by documenting successful accrual, retention, and protocol adherence.

ELIGIBILITY:
Inclusion Criteria:

1. women with a diagnosis of any breast cancer within the last three years
2. being >18 years old
3. having a life expectancy of >12 months
4. report experiencing pain on at least 10 days in the last month and rate their pain in the past week as a 4 or greater on a 0-10 scale. The combination of these items assess patients level of persistent pain (in the last month) and pain severity with an accurate recall period (i.e., last week; >4).

Exclusion Criteria:

1. cognitive impairment as indicated by a baseline Folstein Mini-Mental Status Examination of <2588
2. brain metastases
3. presence of a severe psychiatric condition or a psychiatric condition (e.g., suicidal intent) that would contraindicate safe participation in the study as indicated by the medical chart, treating oncologist, or medical/study staff interactions, or 4) current or past (<6 months) engagement in PCST for cancer.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara J Somers, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three consented participants were lost to follow-up or withdrawn prior to completing the baseline assessment and were not randomized.
Period: Overall Study
Arm/Group | Mobile Health Pain Coping Skills Training (mPCST) | mHealth-Education (mHealth-Ed)
Started | 90 | 87
Completed | 79 | 83
Not Completed | 11 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Health Pain Coping Skills Training (mPCST) | mHealth-Education (mHealth-Ed) | Total
Number analyzed (Participants) | 90 | 87 | 177
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 61 | 115
  >=65 years | 36 | 26 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (12.5) | 59.6 (11.4) | 60.3 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 87 | 177
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 85 | 81 | 166
  Unknown or Not Reported | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 6 | 15
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 27 | 51
  White | 53 | 51 | 104
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Pain Severity as Measured by the Brief Pain Inventory (BPI)
Description: Pain Severity will be assessed using the Brief Pain Inventory (BPI) by asking patients about pain on a scale of 0 = no pain to 10 = pain as bad as you can imagine.
Time Frame: Baseline, post-intervention (up to 10 weeks), 3 months, 6 months
Population: Participants with data collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Health Pain Coping Skills Training (mPCST) | mHealth-Education (mHealth-Ed)
Number analyzed (Participants) | 72 | 77
score on a scale
  Baseline | 4.71 (2.05) | 4.51 (1.84)
  Post-intervention | 3.52 (2.04) | 4.69 (2.32)
  3 months | 3.59 (2.37) | 4.15 (2.40)
  6 months | 3.16 (2.12) | 4.13 (2.58)

2. Primary Outcome: Pain Interference as Measured by the Brief Pain Inventory (BPI)
Description: Pain Interference will be assessed by asking how much pain has interfered with seven daily activities including general activity, walking, work, mood, enjoyment of life, relations with other and sleep within the last 7 days on a scale of 0 = does not interfere to 10 = completely interferes. Reported as the mean score for the seven items.
Time Frame: Baseline, post-intervention (up to 10 weeks), 3 months, 6 months
Population: Participants with data collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Health Pain Coping Skills Training (mPCST) | mHealth-Education (mHealth-Ed)
Number analyzed (Participants) | 72 | 77
score on a scale
  Baseline | 4.64 (2.56) | 4.76 (2.30)
  Post-intervention | 3.28 (2.34) | 4.79 (2.55)
  3 months | 3.22 (2.47) | 4.11 (2.60)
  6 months | 2.92 (2.49) | 4.04 (2.90)

3. Primary Outcome: Change in Fatigue
Description: The Patient Reported Outcomes Measurement Information System (PROMIS) six-item Fatigue Scale is a self-report measure of fatigue symptoms. Items ask patients to evaluate symptoms from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that is likely to decrease one's ability to carry out daily activities. Reported as a T-score with a range of 0 to 100, with a mean score of 50 and a standard deviation of 10. A higher score indicates greater fatigue.
Time Frame: Baseline, post-intervention (up to 10 weeks), 3 months, 6 months
Population: Participants with data collected.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Mobile Health Pain Coping Skills Training (mPCST) | mHealth-Education (mHealth-Ed)
Number analyzed (Participants) | 72 | 77
T-score
  Baseline | 60.60 (7.67) | 60.59 (7.33)
  Post-intervention | 56.38 (8.12) | 58.95 (7.36)
  3 months | 56.34 (8.38) | 58.02 (7.83)
  6 months | 54.25 (8.97) | 58.52 (7.86)

4. Primary Outcome: Physical Disability as Measured by the Patient Care Monitor (PCM)
Description: Physical disability will be assessed using 4-item form Patient Care Monitor (PCM) scale. The four items ask about patients' ability to run, do light physical work or fun activities, do hard physical work or fun activities, and ability to function normally in the last 7 days (0 = not a problem to 10 = as bad as possible). Reported as the mean score for the four items.
Time Frame: Baseline, post-intervention (up to 10 weeks), 3 months, 6 months
Population: Participants with data collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Health Pain Coping Skills Training (mPCST) | mHealth-Education (mHealth-Ed)
Number analyzed (Participants) | 72 | 77
score on a scale
  Baseline | 5.56 (2.45) | 5.87 (2.23)
  Post-intervention | 4.62 (2.40) | 5.64 (2.30)
  3 months | 4.66 (2.67) | 5.29 (2.43)
  6 months | 4.20 (2.77) | 5.31 (2.62)

5. Secondary Outcome: Self-Efficacy for Pain Control as Measured by the Chronic Pain Self-Efficacy Scale
Description: The self-efficacy for pain management will be assessed using 5-item Chronic Pain Self-Efficacy scale. This sub-scale contains 5 items that inquire about patients' certainty about degree of pain control, pain during daily activities, controlling pain during sleep, and making pain reductions without extra medication. These items will be answered on a scale of 10 = very uncertain to 100 = very certain scale and averaged.
Time Frame: Baseline, post-intervention (up to 10 weeks), 3 months, 6 months
Population: Participants with data collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Health Pain Coping Skills Training (mPCST) | mHealth-Education (mHealth-Ed)
Number analyzed (Participants) | 72 | 77
score on a scale
  Baseline | 54.69 (17.79) | 56.09 (18.09)
  Post-intervention | 64.46 (20.42) | 55.12 (18.64)
  3 months | 65.27 (21.58) | 56.60 (18.97)
  6 months | 66.03 (23.17) | 58.49 (23.52)

6. Secondary Outcome: Pain Catastrophizing as Measured by the Coping Strategies Questionnaire
Description: Pain catastrophizing will be assessed with the 6-item pain catastrophizing sub-scale of the Coping Strategies Questionnaire. These items ask about patients' tendency to catastrophize when faced with pain and are answered on a scale of 0 = never to 6 = always and averaged.
Time Frame: Baseline, post-intervention (up to 10 weeks), 3 months, 6 months
Population: Participants with data collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Health Pain Coping Skills Training (mPCST) | mHealth-Education (mHealth-Ed)
Number analyzed (Participants) | 72 | 77
score on a scale
  Baseline | 1.67 (1.41) | 1.83 (1.13)
  Post-intervention | 1.22 (1.05) | 1.60 (1.03)
  3 months | 1.12 (1.06) | 1.53 (1.16)
  6 months | 1.00 (1.12) | 1.60 (1.18)

7. Secondary Outcome: Cost-Effectiveness
Description: We will create a composite cost variable based on patient time, medical resource use, productivity, and the EQ-5D.The EQ-5D is a measure of health status that can be linked to population-based preference weights is widely used in economic evaluations. It is short, assessing 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). The respondent indicates no problems, some problems, or severe problems in each dimension.
Time Frame: Baseline, post intervention(up to 10 weeks or however long the intervention lasts), 3-month and 6- month: approximately 25 minutes each time
Reporting Status: Not Posted, anticipated posting 2026-03

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Mobile Health Pain Coping Skills Training (mPCST) | mHealth-Education (mHealth-Ed)
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/87
Other Adverse Events (participants affected / at risk) | 0/90 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT04175639/Prot_SAP_001.pdf
  • Informed Consent Form (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT04175639/ICF_000.pdf